CLINICAL TRIAL: NCT04876755
Title: An Open Label, Dose Comparison Study to Assess the Efficacy of MBM-02 (Tempol) as a Treatment for Patients Diagnosed With Prostate Cancer in Biochemical Recurrence
Brief Title: MBM-02 (Tempol) for the Treatment of Biochemical Recurrent Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Matrix Biomed, Inc. (Industry)
Collaborators: Prostate Oncology Specialists (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MBI-17-01
Expanded Access: NCT04337099 (Available)
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer Recurrent; Biochemical Recurrent Prostate Cancer
MeSH Terms: interventions — tempol; TEMPOL-H

STUDY DESIGN:
Intervention Model Description: For the dose comparison phase, five entry dosing regimens will be explored and represented by Cohort 1 through Cohort 5.
  The first 3 patients (Cohort 1) will begin with a total daily dose (TDD) of 600 mg of MBM-02.
  The study will employ a 3+3 design with Cohort 5 dose at 1600 mg/day.
  Cohort 6 will enroll up to 40 patients at 1600 mg/day of MBM02.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): Cohort 1 patients will administered 600 mg/day of MBM-02 for 20 weeks.
  Interventions: Drug: MBM-02
- Cohort 2 (Experimental): Cohort 2 patients will administered 1000 mg/day of MBM-02 for 20 weeks.
  Interventions: Drug: MBM-02
- Cohort 3 (Experimental): Cohort 3 patients will administered 1200 mg/day of MBM-02 for 20 weeks.
  Interventions: Drug: MBM-02
- Cohort 4 (Experimental): Cohort 4 patients will administered 600 mg/day of MBM-02 for 20 weeks.
  Interventions: Drug: MBM-02
- Cohort5 (Experimental): Cohort 5 patients will administered 600 mg/day of MBM-02 for 20 weeks.
  Interventions: Drug: MBM-02
- Cohort 6 (Experimental): Cohort 6 patients will administered 600 mg/day of MBM-02 for 20 weeks.
  Interventions: Drug: MBM-02

INTERVENTIONS:
Drug: MBM-02 — MBM-02 is an HIF-1 and HIF-2 inhibitor.
  Other Names: Tempol; 4-hydroxy-tempo; 4-hydroxy-2,2,6,6-tetramethylpiperidine-1-oxyl

SUMMARY:
This is an open label trial to assess the efficacy of MBM-02 (Tempol) as a treatment for patients diagnosed with prostate cancer in biochemical recurrence.

DETAILED DESCRIPTION:
Preliminary data shows MBM-02 has anti-prostate cancer activity without hormone suppression or toxicity to non-cancerous cells and organs.

Solid tumors contain hypoxic regions (low oxygen) due to their high rates of cell proliferation and formation of aberrant blood vessels. Intratumoral hypoxia is associated with increased risk of invasion, metastasis, and patient mortality. Cancer cells respond to hypoxia by stabilizing hypoxia-inducible factor 1 (HIF-1) and hypoxia inducible factor 2 (HIF-2). HIF-1 and HIF-2 activate a transcription of genes encoding proteins that mediate major adaptive responses to hypoxia that are critical for cancer cell survival. Without activation of HIF-1 and HIF-2, cancer cells would not survive.

MBM-02 has been shown to inhibit the genes responsible for prostate carcinogenesis, HIF-1 and HIF-2.

This trial is an open label study that will employ a 3+3 escalation design up to 1600 mg/day. Patients will be exposed to study drug for 20 weeks. PSA and scans will be taken at baseline and week 20 for efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Male 18 years or older;
2. Histologically or cytologically confirmed diagnosis of prostate cancer;
3. Patient must have had previous treatment with definitive surgery or radiation therapy, cryoablation, or brachytherapy;
4. Patient may have prior salvage therapy (surgery, radiation or other local ablative procedures) within 6 months prior to randomization if the intent was for cure. Prophylactic radiotherapy to prevent gynecomastia within 4 weeks prior to randomization is allowed
5. Patient must have evidence of biochemical failure after primary therapy and subsequent progression. Biochemical failure is declared when the PSA reaches a threshold value after primary treatment and it differs for radical prostatectomy or radiation therapy:

   1. For radical prostatectomy the threshold for this study is PSA ≥ 0.8ng/mL
   2. For radiation therapy the threshold is a PSA rise of 2 ng/mL above the nadir PSA achieved post radiation with or without hormone therapy (2006 RTOG-ASTRO Consensus definition).
6. PSA progression requires a PSA rise above the threshold measured at any time point since the threshold was reached;
7. PSA doubling time ≤ 12 months. PSA calculation requires two consecutive PSA rises (PSA2 and PSA3) above the threshold PSA (total 3 PSA values); PSA2 and PSA3 must be obtained within 12 months of study entry. All baseline PSAs should be obtained at the same reference lab.
8. ECOG performance status less than or equal to 2;
9. Ability to swallow the study drugs;
10. If a male with a female partner of child bearing potential, adequate methods of contraception must be employed;
11. If male, no sperm donation for 90 days until after the conclusion of the study;
12. Be properly informed of the nature and risks of the clinical investigation, comply with all clinical investigation-related procedures, and sign an Informed Consent Form prior to entering the clinical investigation;
13. Be able to participate for the full term of the clinical investigation;
14. Have a Karnofsky performance status of >70;
15. Have a life expectancy ≥ 6 months; and
16. Have adequate baseline organ function (hematologic, liver, renal, nutritional and metabolic):

Hematology:

Absolute neutrophil count (ANC) ≥1.5 Hemoglobin ≥ 10 g/dL Platelets ≥ 100,000 per microliter of blood

Hepatic:

Total bilirubin ≤ 2 x ULN Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤2.5 x ULN

Renal:

creatinine clearance (CrCl) ≥ 60 ml/min within 2 weeks prior to registration determined by 24-hour collection or estimated by Cockcroft-Gault formula: CrCl male = [(140 - age) x (wt in kg)] [(Serum Cr mg/dl) x (72)] CrCl female = 0.85 x (CrCl male)

Exclusion Criteria:

1. Evidence of metastatic disease on imaging studies (CT and/or bone scan);
2. Diagnosis of diabetes mellitus defined as:

   1. Fasting blood glucose > 126 mg/dl or,
   2. Random blood glucose > 200 mg/dl
   3. Hemoglobin A1C > 6.5%
3. Patients with QTc >480 msec
4. Need for treatment with any conventional modality for prostate cancer (surgery, radiation therapy, and hormonal therapy);
5. Treatment within the last 30 days with any investigational drug;
6. Radiation therapy within prior 6 months (prophylactic radiotherapy to prevent gynecomastia within 4 weeks prior to randomization is allowed);
7. Patient with previous or concurrent malignancy. Exceptions are made for patients who meet any of the following conditions: Basal cell or squamous cell carcinoma of the skin or prior malignancy that has been adequately treated and patient has been continuously disease free for ≥ 2 years;
8. Evidence of a significant medical illness, or a psychiatric illness/social situation that would, in the investigator's judgment, make the patient inappropriate for this study;
9. Refractory nausea and vomiting, malabsorption, biliary shunt, or significant bowel resection that would preclude adequate absorption of the study drug;
10. Have had a recent, serious, non-malignant medical complication that, in the opinion of the investigator, makes the individual unsuitable for study participation;
11. Have used an investigational drug within 28 days of the initiation of study treatment;
12. Have a history of a positive blood test for HIV;
13. At the time of screening, have a significant active medical illness which, in the opinion of the investigator, would preclude completion of the study; and
14. Body weight less than 35 kg (77 lbs.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 55 (Estimated)
Dates: Start 2021-05-30 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Reduction in Serum PSA | baseline to week 20
  To determine whether the proportion of patients who achieve a ≥ 50% decline in serum PSA after 16 weeks of protocol therapy.

SECONDARY OUTCOMES:
PSA progression | baseline to week 20
  To determine the median time to PSA progression from the start of protocol therapy with MBM-02 among men with biochemically recurrence prostate cancer.
Percent Change in PSA | baseline to week 20
  To determine the mean percent change from baseline after 16 weeks of protocol therapy compared with pre-treatment in PSA doubling time. The pre-treatment PSA doubling time will be determined based upon all PSA measurements obtained within 3 months prior to Day 1 of protocol therapy, with a minimum of three PSA measurements spaced at least 14 days apart

CONTACTS AND LOCATIONS:
Locations (1):
- Prostate Oncology Specialists, Marina del Rey, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thomas R, Sharifi N. SOD mimetics: a novel class of androgen receptor inhibitors that suppresses castration-resistant growth of prostate cancer. Mol Cancer Ther. 2012 Jan;11(1):87-97. doi: 10.1158/1535-7163.MCT-11-0540. Epub 2011 Dec 15. PMID 22172488
- See also: Related Info — http://matrixbiomed.com